CLINICAL TRIAL: NCT03785600
Title: A Sleep Intervention to Improve Rehabilitation in Veterans With Chronic mTBI
Brief Title: Improving Sleep in Veterans With TBI
Acronym: SPTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: D2947-W; IK2RX002947 (NIH)
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; sleep-wake disturbances; Veterans; chronic pain
MeSH Terms: conditions — Brain Injuries, Traumatic; Chronic Pain | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive MBLT or a sham/no-light control. Subjects randomized to receive MBLT will be given a light box (LightPad, Aurora Light Solutions) to take home. Subjects randomized to receive the sham/no-light control will be given a modified negative ion generator.
Who Masked: Participant
Masking Description: Participants will be blinded to the intervention by way of study personnel's description. Subjects will be told that both devices may or may not be active and thus, will be unaware that all light boxes are active and all negative ion generators are inactivated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning Bright Light Therapy (Experimental): Morning bright light: Sitting in front of a lightbox for 60 minutes every morning within 90 minutes of waking up.
  Interventions: Device: Morning Bright Light Therapy
- Negative Ion Generator (Sham Comparator): Negative ion generator: Sitting in front of a modified negative ion generator for 60 min every morning within 90 minutes of waking up.
  Interventions: Device: Negative Ion Generator

INTERVENTIONS:
Device: Morning Bright Light Therapy — Morning bright light: Sitting in front of a lightbox for 60 minutes every morning within 90 minutes of waking up.
  Other Names: Lightbox, light therapy
  Arms: Morning Bright Light Therapy
Device: Negative Ion Generator — Negative ion generator: Sitting in front of a modified negative ion generator for 60 min every morning within 90 minutes of waking up.
  Arms: Negative Ion Generator

SUMMARY:
Traumatic brain injury (TBI) is a major cause of disability in the Veteran population, often resulting in chronic pain and sleep disturbances, among other issues. Extensive rehabilitative efforts are usually required and often prevent return to the workforce and community. Disturbed sleep and excessive daytime sleepiness are among the most pervasive and enduring problems after TBI, which the investigators hypothesize is a significant contributor to these functional impairments and an impediment toward rehabilitation. Thus, this research aims to enhance sleep quality as a means to reduce pain and improve quality of life and functional outcome measures in Veterans with TBI. The investigators predict that the proposed intervention, morning bright light therapy, if found effective, will be cost-effective, rapidly deployable, and highly accepted by Veterans with TBI.

DETAILED DESCRIPTION:
Each year ~2.5 million people sustain a traumatic brain injury (TBI). Also a prominent general public health issue, TBI is particularly prevalent in Veterans, with 60-80% reporting a history of TBI. Over 80% of all TBI are categorized as mild TBI (mTBI), which is associated with a myriad of short- and long-term complications. Two of the principal complicating factors associated with mTBI are sleep-wake disturbances (e.g., insomnia, excessive daytime sleepiness, and circadian rhythm sleep disorders) and chronic pain, including headache and diffuse/global pain. Sleep-wake disturbances and chronic pain have an independent prevalence of ~70%, individually impair quality of life, impede effective rehabilitative therapies, and have staggering functional and economic impacts.

Furthermore, there is a strong bidirectional relationship between sleep-wake disturbances and pain such that impaired sleep exacerbates pain, which leads to greater impairments in sleep and worse pain. This vicious cycle between sleep disturbances and pain, which is a particularly prevalent and detrimental condition in Veterans with chronic mTBI, represents a central challenge precluding effective treatment and ultimately, improving Veteran quality of life. Although there are pharmacological and non-pharmacological therapies for chronic pain, the presence of TBI significantly complicates the effectiveness of these treatment options, and have significant adverse effects (e.g., long-term prescription opioid dependence, misuse, or overdose). The investigators believe there is profound potential to intervene at the sleep level, and, by improving sleep quality, enable Veterans with chronic mTBI to better manage their pain and end this vicious cycle.

This proposal aims to apply a sleep intervention to improve chronic pain in Veterans with mTBI. The investigators propose to use morning bright light therapy (MBLT), a readily deployable, cost-effective, non-pharmacologic, and home-based sleep intervention, to improve sleep-wake disturbances and therefore ameliorate chronic pain and improve quality of life in Veterans with chronic mTBI. Outcomes will be assessed pre- and post-intervention, and at a 3-month follow-up time point. The central hypothesis is that MBLT will improve sleep quality and ameliorate pain, resulting in improved quality of life in Veterans with chronic mTBI.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Medical record-confirmed diagnosis of mTBI
* Current self-reported sleep-wake disturbances

  * defined by clinically abnormal Insomnia Severity Index and/or Functional Outcomes of Sleep scores
* Moderate to severe pain

  * defined as a score of 4 on an 11-point scale94) persisting for longer than 6 months
* English speaking with phone access

Exclusion Criteria:

Exclusion Criteria:

* Decisional impairment and/or dementia
* Current usage of a lightbox or negative ion generator
* Shift work
* History of macular degeneration and/or bipolar disorder
* Evidence for suicidal ideation
* Cancer diagnosis within the past 6 months
* Surgery within the past 6-12 months
* Substance abuse within the past 6-12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan E Elliott, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliott JE, Brewer JS, Keil AT, Ligman BR, Bryant-Ekstrand MD, McBride AA, Powers K, Sicard SJ, Twamley EW, O'Neil ME, Hildebrand AD, Nguyen T, Morasco BJ, Gill JM, Dengler BA, Lim MM. Feasibility and acceptability for LION, a fully remote, randomized clinical trial within the VA for light therapy to improve sleep in Veterans with and without TBI: An MTBI2 sponsored protocol. PLoS One. 2025 Jan 7;20(1):e0305305. doi: 10.1371/journal.pone.0305305. eCollection 2025. PMID 39775195

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morning Bright Light Therapy | Negative Ion Generator
Started | 53 | 24
Completed | 44 | 20
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morning Bright Light Therapy | Negative Ion Generator | Total
Number analyzed (Participants) | 44 | 20 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (13.4) | 51.8 (14.3) | 53.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 34 | 16 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 0 | 7
  Not Hispanic or Latino | 37 | 19 | 56
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 38 | 16 | 54
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Years of Education [Mean (Standard Deviation); unit: years] | 16.5 (1.8) | 15.6 (1.9) | 16.2 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reported Pain
Description: NIH Patient Reported Outcomes Measurement Information System (PROMIS) pain interference short-form 4a.
  4 questions; each question is a 1-5 Likert scale, total score range is 4-20. Higher scores represent greater pain interference.
  *all are reported as total score, no subscale scores present.
Time Frame: Pre- and post-4 weeks of Morning Bright Light Therapy (MBLT) or sham treatment.
Measure: Mean (Standard Deviation); unit: Score on Pain Interference
Arm/Group | Morning Bright Light Therapy | Negative Ion Generator
Number analyzed (Participants) | 44 | 20
Score on Pain Interference
  Mean Pre-Intervention Pain Interference | 9.8 (4.8) | 10.2 (4.7)
  Mean Post-Intervention Pain Interference | 9.3 (4.8) | 10.0 (5.0)
Statistical Analysis 1: Comparison: Morning Bright Light Therapy vs Negative Ion Generator; Test type: Other; p < 0.02, t-test, 2 sided — a priori threshold is <0.05

ADVERSE EVENTS:
Time Frame: Adverse event data was collected started immediately after consent and ended after participants completed all study activities (up to 20 weeks).
Arm/Group | Morning Bright Light Therapy | Negative Ion Generator
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/24
Other Adverse Events (participants affected / at risk) | 0/53 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morning Bright Light Therapy (N=53) | Negative Ion Generator (N=24)
Non-Serious (Psychiatric disorders) | 0 (0) | 1 (1) — Subject reported anxiety from dark adaptation of Dim Light Melatonin Onset saliva protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03785600/Prot_001.pdf
  • Informed Consent Form (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03785600/ICF_000.pdf